CLINICAL TRIAL: NCT05717842
Title: Simultaneous Prospective Kidney Transplant Assessment in Combined Liver Kidney
Brief Title: Simultaneous Prospective Kidney Transplant Assessment in Combined Liver Kidney Candidates
Acronym: RECOVERY
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Jerome A. Josephs Fund for Transplant Innovation Fund (Unknown)
Responsible Party: Principal Investigator, Muhammad Yahya Jan, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: 15853
Record Dates: First submitted 2022-12-02; First posted 2023-02-08 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Transplant
Keywords: Liver; Kidney

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with ESLD and eGFR between >=25 and <=40ml/min: 1. > 18 years old
  2. Listed for Liver Transplant for ESLD and Kidney Transplant (not on dialysis)
  3. Candidates with two native kidneys.
  4. Willing to participate and sign informed consent
  Interventions: Radiation: Nuclear Medicine Scan

INTERVENTIONS:
Radiation: Nuclear Medicine Scan — Mercaptoacetyltriglycine 3 (Mag 3) Nuclear Medicine Scan

SUMMARY:
The purpose of the study is to determine how much a persons kidney function recovers after receiving a simultaneous liver kidney transplant. The investigators will be contacting patients with kidney dysfunction with estimated GFR between 25 and 40 (not on dialysis treatment) who are listed to receive a simultaneous liver kidney (SLK) transplant to look at this function recovery. The investigators hope to develop a criteria based on GFR measurement, kidney function calculations from native kidneys vs transplanted kidney and compare the contributions, and correlate with estimated GFR on basic metabolic panel (BMP: a blood test) to predict higher chances of recovery of native kidney function.

DETAILED DESCRIPTION:
Study design

Study will be a pilot longitudinal prospective study. SLK transplant listed patients will be recruited from the outpatient Liver Kidney Transplant Clinic at Medical Diagnostic Clinic (MDC) as well as inpatients admitted to IU University Hospital. Listing status for SLK transplant will be confirmed and patients will be scheduled for a Mag3 nuclear medicine scan at IU University Department of Nuclear medicine. For study purposes, this scan will be done pre and post-transplant to compare the results.

Methods:

Inclusion/Exclusion criteria:

Inclusion:

1. > 18 years old
2. Listed for Liver Transplant for ESLD and Kidney Transplant based on eGFR ranging from ≥ 25 to ≤40 mL/min/1.73m2 (not on dialysis at time of surgery)
3. Candidates with two native kidneys.
4. Willing to participate and sign informed consent form.

Exclusion Criteria:

1. Unstable patients (e.g. in the ICU or those who are on Continous Renal Replacement Therapy (CRRT) who cannot complete the nuclear medicine scan or those on Hemodialysis
2. Prior history of any solid organ transplant.
3. Those who are currently pregnant or breast feeding.
4. Patients with a history of Adult Polycystic Kidney Disease

Data collection: Data collection will be done in RedCap©️ These data forms will incorporate a comprehensive list of variables:

1. Participants demographics and BMI
2. Reason for ESLD and complications listed in Medical Chart
3. Medication list
4. Results of Nuclear medicine scan, eGFR on Basic Metabolic Panel, measurement of eGFR by Cystatin C, 24 hour urinary creatinine clearance and measurement of urinary NGAL level. Radiographically: kidney size, presence of findings such as cysts, stones etc.
5. Post SLK transplant complications including need for Dialysis, delayed graft function, episodes of rejection, infections and any reason for admission to the hospital
6. Adherent to Immunosuppression regimen, and type of Immunosuppression regimen
7. BP readings at follow up clinic visits
8. Any post SLK transplant imaging for kidney size and any findings (if any imaging is performed for any other indication, none will done for the research study).

Participants will be informed about the results of their studies. Participation will be voluntary. Compensation will be provided once in the form of $25 gift card that will be provided upon completing participation for the nuclear medicine scan 10 months after patients receive their SLK transplant. Patients and their insurance will not be charged and the testing will be invoiced to the study grant.

Provisions for post-study care No provision will be provided for care regarding incidental findings on the nuclear medicine scan. They will be given information regarding referral to seeking appropriate care. No expenses will be reimbursed for this care.

Participant timeline:

Enrollment of participants will be done starting February 2023 and completed by December 2023

Statistical Analyses:

Sample size:

Estimated number of participants is determined by participants listed for SLK transplant. An estimated 15 participants are planned to be recruited. As this is a pilot study, all participants at IU will be asked to participate with a future goal of a multi-center study.

Plans for assessment and collection of outcomes:

Data will be collected in IU RedCap registry, which is a secure platform. Data will be entered in Redcap, coded, secured, and stored. Any raw data collection (source documents) will be kept in a locked cabinet in a locked office. Data will be processed with SPSS data management software.

Confidentiality Information about potential and enrolled participants will be collected, shared, and maintained in a manner that protects confidentiality before, during, and after the study.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old
2. Listed for Liver Transplant for ESLD and Kidney Transplant (not on dialysis at time of transplant surgery)
3. Candidates with two native kidneys.
4. Willing to participate and sign informed consent form.

Exclusion Criteria:

1. Unstable patients (e.g. in the ICU or those who are on Continuous Renal Replacement Therapy (CRRT) who cannot complete the nuclear medicine scan or those with AKI on Hemodialysis
2. Prior history of any solid organ transplant.
3. Those who are currently pregnant or breast feeding.
4. Patients who have Autosomal Dominant polycystic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have end stage liver disease (ESLD) and kidney dysfunction, who are not on dialysis and have eGFR >=25 and <=40 ml/min for a duration of at least 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
perform a nuclear medicine scan prior to SLK transplant | up to 100 weeks
  To determine split kidney function with a Mag3 (Mercaptoacetyltriglycine 3) nuclear medicine renal scan as part of the study procedures.

SECONDARY OUTCOMES:
To measure and correlate Clinical, laboratory and Radiographic data at the time of SLK transplant will be reviewed | up to 100 weeks
  This includes standard testing performed at our center prior to SLK transplant which are standard of care. This will include measurement of eGFR by Cystatin C.

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No